CLINICAL TRIAL: NCT03321838
Title: Pilot Study of Office Based Vergence and Accommodative Therapy as Treatment of Intermittent Exotropia
Brief Title: Office Based Vergence and Accommodative Therapy and Intermittent Exotropia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiang Chen, Associate clinical professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XT1
Record Dates: First submitted 2017-10-15; First posted 2017-10-26 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Intermittent Exotropia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accommodative/vergence therapy (Experimental): Accommodative/vergence therapy (60 minutes per visit, one time per week, 12-14 weeks) and home reinforcement (15 minutes each time, five times per week, 12-14 weeks) will be provided to patients of treatment group. These therapy includes accommodative, vergence and anti-suppression technique. No drug is used during the whole therapy process.
  Interventions: Behavioral: accommodative/vergence therapy

INTERVENTIONS:
Behavioral: accommodative/vergence therapy — Accommodative/vergence therapy (60 minutes per visit, one time per week, 12-14 weeks) and home reinforcement (15 minutes each time, five times per week, 12-14 weeks) will be provided to patients of treatment group. These therapy includes accommodative, vergence and anti-suppression technique. No drug is used during the whole therapy process.

SUMMARY:
This pilot study is designed specifically to determine the short-term effect of OBVAT on intermittent exotropia in terms of 4 key areas (Standardizing reported outcomes of surgery for intermittent exotropia): control score, alignment, near stereoacuity and quality of life score. Result of this pilot study will be used to determine whether a full-scale RCT should be conducted to evaluate the short and long term effectiveness of OBVAT.

DETAILED DESCRIPTION:
All enrolled px received 16-20 sessions of OBVAT, 60 minutes per visit, one time per week; Home reinforcement, 15 minutes each time, five times per week.

1. Primary outcome measure： A. Change in the office based intermittent exotropia control score
2. Secondary outcome measures A. Change in Look And Cover, then Ten seconds of Observation Scale for Exotropia (LACTOSE) B. Change in Newcastle Control Score (NCS) C. Change in Chinese intermittent exotropia questionnaire (CIXTQ) D. Change in near stereopsis by Preschool randot near stereoacuity E. Change in size of distant deviation angle by prism alternating cover test F. Change in size of near deviation angle by prism alternating cover test

ELIGIBILITY:
Inclusion Criteria:

1. 8 to 18 years old
2. deviation meeting all of the following criteria: A. intermittent or constant exotropia at distance (mean of 3 baseline assessments of distance control> or = Grade 2) B. intermittent exotropia at near (at least 1 of 3 assessments of near control at the baseline visit Grade 2-4) C. distance and near exodeviation both between 15 to 35 prism diopters (PD) measured by prism and alternate cover test (PACT); D. near deviation not exceeding the distance deviation by >10PD by PACT (i.e., convergence insufficiency type IXT excluded)
3. cycloplegic objective refraction spherical equivalent (SE) refractive error between -6.00 diopters (D)and +1.00 D inclusive in either eye
4. Patients must be wearing the updated refractive correction (spectacles or contact lenses) for at least 1 week if refractive error (based on cycloplegic refraction performed within 6 months) meets any of the following:

   A. Myopia >-0.50 D spherical equivalent in either eye B. Anisometropia >1.00 D spherical equivalent C. Astigmatism in either eye >1.50 D
5. Refractive correction must meet the following guidelines:

   A. Anisometropia spherical equivalent must be within 0.25 D of the full anisometropic difference B. Astigmatism cylinder must be within 0.25 D of full correction and axis must be within 5 degree C. For hyperopia and myopia, the spherical component can be reduced by investigator discretion provided reduction is symmetrical and results in residual (i.e., uncorrected) spherical equivalent refractive error that does not exceed +1.50 D spherical equivalent hyperopia or -0.50 D spherical equivalent myopia
6. Gestational age >34 weeks
7. Birth weight >1500 g
8. No previous surgical or nonsurgical treatment for IXT other than single vision refractive correction (e.g. PALs, Bifocals, patching, or deliberate over-minus with spectacles more than 0.50 D)
9. No vision therapy or orthoptics for any reason within the last year
10. No prior strabismus surgery or botulinum injection, intraocular surgery, or refractive surgery
11. No strabismus surgery planned
12. vision correctable to at least 20/25 or better at distance and near in each eye.
13. Px needs to have a computer at home which can connect to internet

Exclusion Criteria:

1. Patient with nystagmus, restrictive or paretic strabismus
2. Patient with amblyopia, which is defined as >or = 0.2 logarithm of the minimum angle of resolution units of interocular difference and > or = 0.3 logarithm of the minimum angle of resolution units in one eye ( Variability of stereoacuity in intermittent exotropia)
3. Regular use of any ocular or systemic medications known to affect accommodation or vergence system, such as atropine, pirenzepine, and anti-epileptic medications in recent 3 months；
4. developmental disability, attention deficit hyperactivity disorder(ADHD), or learning disability diagnosis in children that in the investigator's discretion would interfere with office-based treatment；
5. Relocation anticipated for 2 years；
6. Significant ocular or neurologic disorders (e.g. cerebral palsy) other than strabismus
7. Vertical deviation greater than 1 pd in cover test
8. Household member already in the study.
9. Any eye care professional, ophthalmic technician, medical student, or optometry student

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Office based intermittent exotropia control score | Baseline visit, 7th visit(7 weeks after BL), 15th visit (15 weeks after BL)
  Office based intermittent exotropia control score is an office based score to assess the control of intermittent exotropia. Minimum score is 0 (best score, phoria) and Maximum score is 5(worst score, constant tropia). Change in Office based intermittent exotropia control score after 14 weeks of vision therapy

SECONDARY OUTCOMES:
Look And Cover, then Ten seconds of Observation Scale for Exotropia(LACTOSE) | Baseline visit, 7th visit(7 weeks after BL), 15th visit (15 weeks after BL)
  Look And Cover, then Ten seconds of Observation Scale for Exotropia (LACTOSE) is an office based score to assess the control of intermittent exotropia. Minimum score is 0 (best score, phoria) and Maximum score is 4(worst score, constant tropia). Change in score after 14 weeks of vision therapy.
Newcastle Control Score | Baseline visit, 7th visit(7 weeks after BL), 15th visit (15 weeks after BL)
  Newcastle Control Score is an office based and home based score to assess the control of intermittent exotropia. Minimum score is 0 (best score) and Maximum score is 6(worst score). Change in score after 14 weeks of vision therapy.Change in score after 14 weeks of vision therapy.
Chinese intermittent exotropia questionnaire | Baseline visit, 7th visit(7 weeks after BL), 15th visit (15 weeks after BL)
  Change in Chinese intermittent exotropia questionnaire after 14 weeks of vision therapy.
Preschool randot near stereoacuity | Baseline visit, 7th visit(7 weeks after BL), 15th visit (15 weeks after BL)
  Change in near stereopsis by Preschool randot near stereoacuity after 14 weeks of vision therapy.
deviation angle | Baseline visit, 7th visit(7 weeks after BL), 15th visit (15 weeks after BL)
  Change in size of distant deviation angle by prism alternating cover test after 14 weeks of vision therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Chen xiang, Study Director — associate chief physician
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ma MM, Kang Y, Scheiman M, Chen X. Office-based Vergence and Accommodative Therapy for the Treatment of Intermittent Exotropia: A Pilot Study. Optom Vis Sci. 2019 Dec;96(12):925-933. doi: 10.1097/OPX.0000000000001454. PMID 31834152